CLINICAL TRIAL: NCT03517046
Title: A Multi-center, Open-label, Phase I Trial to Assess the Safety for Treatment of Autologous Chondrocytes Implantation With CartiLife for Patients With Chondral Defects in the Knee
Brief Title: Study to Assess the Safety of Treatment of Articular Cartilage Lesions With CartiLife®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biosolution Co., Ltd. (Industry)
Collaborators: Kyung Hee University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCTT-CTL-I
Record Dates: First submitted 2018-03-08; First posted 2018-05-07 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-03

CONDITIONS: Articular Cartilage Lesion of Knee
Keywords: Arthritis; Articular Cartilage; Autologous Chondrocyte Implantation; Degenerative Arthritis; Cartilage Lesion; Cartilage Defect
MeSH Terms: conditions — Arthritis; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CartiLife (low-dose group) (Experimental): Total defect volume in low-dose group is less than 2 ㎤. Low- and high-dose group are sequentially processed.
  Interventions: Drug: CartiLife
- CartiLife (high-dose group) (Experimental): Total defect volume in High-dose group is 2 ~ 4 ㎤.
  Interventions: Drug: CartiLife

INTERVENTIONS:
Drug: CartiLife — Biological: CartiLife® Procedure: CartiLife® is beads (1.0 to 1.5 mm in diameter) in suspension, developed from autologous chondrocytes. The beads are implanted in a volume of 1 cm3 per the capacity of the syringe to the affected area through injection with a fibrin adhesive through minimal arthrotomy.

SUMMARY:
The purpose of this study is to assess the safety and efficacy of implanting bead-type autologous chondrocytes (CartiLife®) obtained by culturing expanded costal chondrocytes of the patient with a chondral defect in the knee. The patients will be assessed clinically using clinical, biochemical and IKDC (International Knee Documentation Committee) outcomes preoperatively as well as 4, 8, 24 and 48 weeks postoperatively to assess the relief of symptoms and joint function.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 19 years old
* Defect size: 2 to 10 ㎠ on the unilateral knee cartilage (up to 4 ㎤ in volume)
* Defect: isolated ICRS (International Cartilage Repair Society) grade III or IV single defect chondral lesion on articular cartilage
* The joint space is maintained over 50% relative to baseline
* Patients that are able to walk without aid
* Patients that agree to abide by strict rehabilitation protocols and follow-up programs
* Patients who provide written consent to the participation of the clinical trial

Exclusion Criteria:

* Patients with inflammatory articular diseases such as rheumatoid arthritis or gouty arthritis
* Patients with arthritis associated with autoimmune disease
* Patients hypersensitive to bovine protein
* Patients with Haemophilia or markedly reduced immune function
* Patients hypersensitive to antibiotics such as gentamicin
* Patients with arterial bleeding and severe venous bleeding
* Patients with other diseases including tumors except for cartilaginous defects of joints
* Patients with a history of radiation treatment and chemotherapy within the past two years
* Patients who are pregnant, nursing a baby or likely to get pregnant
* Patients who participate in concurrent clinical trials or previous clinical trials within 30 days of administration
* Other cases where the investigator deems the patient ineligible for participation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-07-17 (Actual); Primary Completion 2013-12-10 (Actual); Study Completion 2013-12-10 (Actual)

PRIMARY OUTCOMES:
Adverse events | 48 weeks
  Number of adverse events

SECONDARY OUTCOMES:
IKDC (International Knee Documentation Committee) | Baseline to 48 weeks
  Changes in IKDC scores during each visit
  The IKDC Score is a subjective questionnaire filled out by the patient ranges from 0-100, where a score of 100 is interpreted to mean no limitation with sporting activities or daily living and the complete absence of symptoms
X-ray | Baseline 48 weeks
  Changes in structure during each visit

CONTACTS AND LOCATIONS:
Overall Officials: Kyoung Ho Yoon, MD, PhD, Principal Investigator — Kyunghee University Medical Center

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yoon KH, Park JY, Lee JY, Lee E, Lee J, Kim SG. Costal Chondrocyte-Derived Pellet-Type Autologous Chondrocyte Implantation for Treatment of Articular Cartilage Defect. Am J Sports Med. 2020 Apr;48(5):1236-1245. doi: 10.1177/0363546520905565. Epub 2020 Mar 3. PMID 32125878